CLINICAL TRIAL: NCT05300321
Title: Efficacy of Defocus Incorporated Multiple Segments (DIMS) Lens Chinese Myopic Children
Brief Title: DIMS-myopia Progression ADN Axial Length Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY201902
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Myopia, Progressive
Keywords: myopia; axial length; DIMS
MeSH Terms: conditions — Myopia, Degenerative; Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Vision Lens (Experimental): The sunbjects were randomized to allocate in single vision lens group.
  Interventions: Device: frame lens
- Defocus Incorporated Multiple Segments (DIMS) Lens (Experimental): The sunbjects were randomized to allocate in Defocus Incorporated Multiple Segments (DIMS) Lens group.
  Interventions: Device: frame lens

INTERVENTIONS:
Device: frame lens — The subjects were randomized to allocate in Single Vision (SV) lens or Defocus Incorporated Multiple Segments (DIMS) Lens group.

SUMMARY:
To confirm the efficacy of DIMS lenses in controlling myopia progression, we planned a prospective randomized controlled clinical study.

DETAILED DESCRIPTION:
The subjects were randomly assigned into two groups: the control group (SV) and the experimental group (DIMS). The clinical trial assistant took the glasses before examination and returned them after examiners had performed all tests. Examiners were unaware of the spectacle type until the end of the follow-up period. However, the lens type was known by children and parents since the unique appearance of the DIMS lens.

The subjects were provided details about the study design and methodology and their rights as subjects at first visit. We conducted visual acuity tests, subjective and objective refraction measurements, AL measurements, heterophoria at distance and near, and accommodation after obtaining written informed consent from them and their parent.

We conducted follow-up examinations 6 and 12 months after the first visit. In the follow-up examinations, we measured all the examination as do ate the firt visit.

Either the VA with the current spectacles dropped to < 0.8(20/20) or SE of cycloplegic subjective refraction increased ≤-0.50D, the lens power of the spectacles was replaced on the basis of the cycloplegic subjective refraction.

ELIGIBILITY:
Inclusion Criteria:

* The subjects had spherical RE of -1.00 to -6.50 D, astigmatism ≤ 4.00 D, anisometropia ≤ 1.50 D
* Best corrected visual acuity (BCVA) equal to or better than logMAR 0.0 (20/20) in both eyes.

Exclusion Criteria:

* Candidate subjects were excluded from the study if they had strabismus, ocular limitations, or systemic abnormalities affecting vision and ocular motility.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Cycloplegic objective refraction | 12months
  Cycloplegic objective refraction was measured with an autorefractor (Topcon KR8900, Japan).

SECONDARY OUTCOMES:
Axial Length | 12months
  Axial length (AL) was measured with an AL-Scan optical biometer (Nidek, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoqin Chen, MD, Principal Investigator — Tianjin Eye Hospital
Locations (1):
- Tianjin Eye Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No